CLINICAL TRIAL: NCT00180609
Title: Scandinavian Automatic Capture Study
Brief Title: SCANCAP Scandinavian Automatic Capture Study
Status: Completed | Type: Observational
Sponsor: Guidant Corporation (Industry)
Other Study IDs: SCANCAP-1003
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: Automatic threshold test in Insignia Pacemakers from Guidant

SUMMARY:
The primary objective of this study is to document the success rate of the automatic threshold testat pre-discharge in a normal pacemaker patient population implanted with Guidant Insignia Ultra or AVT .

DETAILED DESCRIPTION:
Currently the optimal programming of the pacemaker output considers both pacemaker efficiency (prolonging battery longevity) and patient safety (adequate safety margin). A decrease in the programmed output can be used to increase the projected battery life or to eliminate diaphragmatic or pectoral muscle stimulation. An increase in programmed output may be required to account for increasing thresholds after lead implantation. The ability of an implanted pacemaker to automatically adjust the ventricular output above the pacing threshold while maintaining the appropriate safety margin has been explored since the early 1970s. The Automatic capture feature in the INSIGNIA I Ultra/AVT pacemaker automatically adapts the ventricular pacing output to ensure capture of the ventricle while optimizing the output voltage. The primary objective of this study is to document the success rate of the automatic threshold test in a normal pacemaker patient population by following normal pacemaker follow-up results for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Suitable candidate for a INSIGNIA I Ultra or Insignia I AVT pacemaker (with a ventricular lead). Availability for follow-up at the centre. Willingness to participate in this study. Age 18 or above, or of legal age to give informed consent as specified by national law.

Exclusion Criteria:

* Inability or refusal to sign the Patient Informed Consent. Known pregnancy. Presence of mechanical tricuspid valve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203
Dates: Start 2003-12; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Per D Christensen, MD, Principal Investigator — Medicinsk Afdeling, Sygehus Viborg, Viborg, Denmark
Locations (1):
- Medicinsk Afdeling, Sygehus Viborg, Viborg, Denmark